CLINICAL TRIAL: NCT04888221
Title: Efficacy of Tocilizumab in Association to Steroids in Giant Cell Arteritis With Cerebro-vascular Involvement (ToGiAC)
Brief Title: Efficacy of Tocilizumab in Association to Steroids in Giant Cell Arteritis With Cerebro-vascular Involvement
Acronym: TOGIAC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Roche Chugai (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP191062; 2020-000080-23 (EudraCT Number)
Record Dates: First submitted 2021-03-25; First posted 2021-05-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Giant Cell Arteritis; Neurovascular Disorder
Keywords: Giant Cell Arteritis; ischemic complication/ ischemic event; Cerebro-vascular involvement; Steroids; Tocilizumab; Horton's Giant Cell Arteritis; Vascular Diseases; Neurovascular Diseases; Cerebrovascular Disorders
MeSH Terms: conditions — Giant Cell Arteritis; Vascular Diseases; Cerebrovascular Disorders | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tocilizumab 162mg/0.9mL administered subcutaneously (SC) weekly during 24 weeks (Experimental): Tocilizumab 162mg/0.9mL administered subcutaneously (SC) weekly during 24 weeks
  Interventions: Drug: Tocilizumab
- placebo administered subcutaneously (SC) weekly during 24 weeks (Placebo Comparator): Placebo administered subcutaneously (SC) weekly during 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be administered subcutaneously at a dose of 162mg/0.9mL weekly (each week, on the same day) from week 0 to week 24.
  At the first injection (Baseline D0), a therapeutic education is provided for patients/caregivers who can carry out the injections themselves as part of their usual care.
  Other Names: RoActemra; Actemra
  Arms: tocilizumab 162mg/0.9mL administered subcutaneously (SC) weekly during 24 weeks
Drug: Placebo — Placebo administered subcutaneously (SC) weekly during 24 weeks
  Arms: placebo administered subcutaneously (SC) weekly during 24 weeks

SUMMARY:
A French multicenter randomised and placebo-controlled study recruiting patients who present neurovascular involvement related to GCA (> 60 years) with symptomatic (stroke) or asymptomatic forms. The aim of this study is to assess the efficacy of tocilizumab to induce complete remission of GCA with cerebrovascular involvement (clinical and biological) and absence of clinical and MRI ischemic stroke recurrence at 24 weeks.

DETAILED DESCRIPTION:
Giant cell arteritis (GCA) in the elderly is considered a medical emergency in case of ischemic complication, urgent treatment is needed and high doses of intravenous steroids are used. To date, usual treatments added to steroids have not been shown to be effective in reducing the risk of ischemic event recurrence in GCA.

Recently, the efficacy of tocilizumab has been demonstrated as a steroid-sparing agent and a long-term complete remission agent. The aim of this study is to address the potential benefits of tocilizumab as induction therapy in combination with high dose steroids to improve the neurovascular involvement in GCA.

The study will enroll 66 subjects with GCA (according to ACR criteria or positive temporal artery biopsy) and neurovascular involvement (symptomatic or asymptomatic). It consist of a screening phase (up to 30 days), a baseline/randomization phase and a treatment phase with experimental treatment or placebo (weekly administrated) which could be combined with usual treatments for stroke as antiaggregants and/or anticoagulants (24 weeks). Regular visit will be performed to follow the GCA remission, adverse treatments effects and proceed to radiological and biological evaluations (visit assessment at weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36) until end of study visit at week 52.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Diagnosis of
* GCA (according to ACR criteria or positive temporal artery biopsy) (de novo and/or relapse) And neurovascular involvement:
* Either Ischemic stroke (including TIA) in the vertebro-basilar or carotid territory (symptomatic arterial involvement)
* Either PET uptake of vertebral and/or carotid arteries (extra or intra cranial) and/or angioCT or angioMRI showing arterial involvement consistent with vasculitis (asymptomatic arterial involvement)
* Inclusion should be done
* within 4 weeks after the stroke concerning the "symptomatic" patients
* within 4 weeks after the diagnosis of GCA (or relapse) concerning the patients with asymptomatic neurovascular involvement.
* Within 21 days after starting the corticosteroids
* Signed Informed Consent Form
* Affiliation to social security

Exclusion Criteria:

* Other proven cause of stroke: atrial fibrillation, significant atheromatous stenosis of carotid or vertebro-basilar arteries
* Contraindication to and precaution in use of tocilizumab:

  * Treatment with any investigational agent within 12 weeks (or 5 half-lives of the investigational drug, whichever was longer) of screening
  * Previous treatment with cell-depleting therapies, including investigational agents,including but not limited to Campath (alemtuzumab), anti-CD4, anti-CD5, anti-CD3, anti-CD19, and anti-CD20 within 6 months before the baseline
  * Treatment with IV gamma globulin or plasmapheresis within 24 weeks of baseline
  * Previous treatment with alkylating agents, such as chlorambucil, or with total lymphoid irradiation within 2 months before the baseline
  * Previous treatment with TCZ within 6 months before the baseline
  * Immunization with a live/attenuated vaccine within 4 weeks prior to baseline or simultaneously with tocilizumab treatment
  * Treatment with hydroxychloroquine, cyclosporine A, azathioprine, or mycophenolate mofetil (MMF) within 4 weeks of baseline
  * Treatment with etanercept within 2 weeks; infliximab, certolizumab, golimumab,abatacept, or adalimumab within 8 weeks; or anakinra within 1 week of baseline
  * Previous treatment with tofacitinib within 2 months before the baseline
  * Treatment with cyclophosphamide within 24 weeks of baseline
  * History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies or to prednisone
  * Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (including uncontrolled diabetes mellitus), psychiatric, osteoporosis/osteomalacia, glaucoma, corneal ulcers/injuries, or gastrointestinal disease
  * Current liver disease, as determined by the investigator
  * History of diverticulitis, diverticulosis requiring antibiotic treatment, or chronic ulcerative lower GI disease such as Crohn's disease, ulcerative colitis, or other symptomatic lower GI conditions that might predispose a patient to perforations
  * Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections (including but not limited to tuberculosis [TB] and atypical mycobacterial disease, hepatitis B and C, and herpes zoster, but excluding fungal infections of the nail beds)
  * Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks of screening
  * Active TB requiring treatment within the previous 3 years
  * Patients treated for TB with no recurrence within 3 years and patients treated for latent TB within 3 years were eligible.
  * Primary or secondary immunodeficiency (history of or currently active)
  * Evidence of malignant disease or malignancies diagnosed within the previous 5 years (except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that had been excised and cured)
  * History of alcohol, drug, or chemical abuse within 1 year prior to screening
  * Body weight >150 kg
  * Serum creatinine >1.4 mg/dL (124 µmol/L) in female patients and 1.6 mg/dL (141 µmol/L) in male patients
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)× 3 Upper limit of normal (ULN)>
  * Platelet count < 100 109/L (100,000/mm3)
  * Hemoglobin < 85 g/L (8.5 g/dL; 5.3 mmol/L)
  * White blood cells <3.0 x109/L (3000/mm3)
  * Absolute neutrophil count < 2.0 x 109/L (2000/mm3)
  * Absolute lymphocyte count < 0.5 X 109/L (500/mm3)
  * Positive hepatitis B surface antigen or hepatitis C antibody
  * Contraindication to aspirin, clopidogrel, steroids use, rifampicin and/or isoniazid
  * Major surgery within 8 weeks prior to screening or planned major surgery within 12 months after randomization, except arterial thrombectomy if necessary for ischemic stroke
  * Transplanted organs (except corneal transplant performed more than 3 months prior to screening)
  * Inability to provide informed consent
  * Participation in another interventional research

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-08-13 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in complete remission of GCA with absence of ischemic stroke recurrence at 24 weeks under tocilizumab. | From date of treatment initiation until 24 weeks.
  Percentage of participants with complete remission of GCA, defined as an absence of clinical signs of GCA, a CRP levels less than 10 mg/l and an absence of new ischemic stroke signs at MRI realized at 24 weeks after the tocilizumab initiation

SECONDARY OUTCOMES:
Compare within tocilizumab and placebo groups the percentage of clinical and MRI ischemic stroke recurrence at 24 weeks | at week 4, 12, 24 and 52.
  the efficacy of weekly tocilizumab on the prevention of stroke recurrence will be measured by the percentage of stroke recurrence compared to control group in patients with GCA during 52 weeks at week 4, 12, 24 and 52
The relapse-free survival | up to 52 weeks
  Number of patients who had relapsed as defined as major if clinical symptoms are present, or as minor in the case of isolated acute pase reactants increase
Compare within tocilizumab and placebo groups the time to remission in patients with GCA during 52 weeks. | at week 4, 12, 24 and 52.
  the time to remission will be assessed in comparison with the control group in patients with GCA during 52 weeks at week 4, 12, 24 and 52 Number of days between treatment induction and signs of remission.
Compare within tocilizumab and placebo groups the improvement of neurovascular radiological involvement during 52 weeks | at week 4, 12, 24 and 52.
  Proportion of patient with neurovascular radiological involvement defined as angio-CT improvement of vasculitis lesions and /or improvement or disappearance of PET FDG uptake.
Compare within tocilizumab and placebo groups the steroid sparing effect at 24 weeks | up to 24 weeks
  Cumulative steroid dose at 24 weeks
Mortality at week 4, 12, 24 and 52 | at week 4, 12, 24 and 52
  Percentages of deaths at week 4, 12, 24 and 52.
Evolution of degree of disability or dependence at week 4, 12, 24 and 52 | at week 4, 12, 24 and 52.
  Percentages of patients with rankin score 0-1
Percentage of Participants with Adverse Events/ serious adverse events | at week 4, 12, 24 and 52.
  Percentage of participants with adverse events, treatment-related adverse events or serious adverse event as assessed by CTCAE v4.0, at week 4, 12, 24 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Sonia ALAMOWITCH, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Saint Antoine Hospital, Neurology Unit, Assistance Publique-Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided